CLINICAL TRIAL: NCT04173546
Title: Systematic Screening and Identification of Psychoactive Substances Users in Young Adults (16 to 25 Years Old) Visiting the Emergency Department
Brief Title: Identification of Psychoactive Substance Users in Young Adults (16 to 25 Years Old) Visiting the Emergency Department
Acronym: DRUGS
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL18_0974
Record Dates: First submitted 2019-11-15; First posted 2019-11-22 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Psychiatric Emergency; Drug Use

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urinary strips will determine the recent consumptions (from a few days to a few weeks according to the products) of seven psychoactive substances (alcohol, tobacco, cannabis, ecstasy, amphetamines, cocaine, morphinics). The detection of some substances in urine works via measurement of the decomposition products from metabolism: cotinine for tobacco, ethyl glucuronide for alcohol, benzoylecgonine for cocaine. Regarding ecstasy, amphetamines, cannabis and morphinics, the detection is done directly in urines. There are seven reading windows (one for each substance) on the Drug Screen: if a colored strip appears in the reading window it means that the detection is negative, otherwise if there is no strip it is considered as positive
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Adolescence is a time for great physical and psychological change and it's often at that period of life that first use of psychoactive substances occurs. Although addiction is rare in teenagers, psychoactive substances abuse can have serious long-term health consequences on them. This is therefore a priority for all healthcare providers to identify early use and abuse of drugs in the youth's population.

The addictive process underlies environmental, genetic and individual causes. That is why it is somehow possible to identify individuals at risk based on some common sociological, cultural and environmental risk factors.

Due to the acute consequences of psychoactive substances abuses, Emergency Departments are main checkpoints for the screening of young drug users. Indeed, one patient out of five admitted in an Emergency Department shows a positive blood alcohol concentration regardless of the reason for their admission. This rate is twice as high as in the overall population. Hence, Emergency Departments are at the front-line for screening, caring, referral and transfer of psychoactive substances users. That is why the Emergency Department is the best place for this study.

In 2004, the special consultations of young consumers were founded in order to deal with these special cases where dependence is not yet established or installed and care has to be adapted to the age. Offering help to this age range represents a real challenge since only 20% of the teenagers come to visit this special consultations on their own initiative. The rest of teenagers are either obliged by their parents or sentenced by a court. The investigators assume that the repetition of care offered to the teenagers by repeated emergency admissions could trigger their own desire to overcome their drug use disorders and visit the Addictionology Department.

ELIGIBILITY:
Inclusion Criteria:

* All patients aged 16 to 25 admitted at the Medical and Psychiatric Emergency Department.
* For adults: those who will agree to participate in this study
* For Minors from the age of 16: those who will agree to participate and want to exercise their rights by themselves or for whom one parent or legal guardian agrees for their participation.

Exclusion Criteria:

* patient who doesn't understand French
* patient under legal protection measures or guardianship
* confused person (GSC < 15)

Ages: 16 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Young people aged 16-25 inclusive, admitted to the Medical and Psychiatric Emergency Department (Building N) of the Edouard Herriot Hospital.
Sampling Method: Probability Sample
Enrollment: 459 (Actual)
Dates: Start 2020-02-11 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2021-04-15 (Actual)

PRIMARY OUTCOMES:
Consumption questionnaire and urinary strips to detect psychoactive substances users | Follow-up time: 3 months
  The primary objective of the study is to evaluate the prevalence of psychoactive substances use among young adults, aged 16 to 25, visiting the Emergency Department.
  This evaluation will be twofold:
  * declarative through a consumption questionnaire (response by Yes or No without score) (whole life, past three months and previous month)
  * analytical by means of a urinary screening for recent consumptions (from a few days to a few weeks according to the products) of seven psychoactive substances (Alcohol, tobacco, cannabis, ecstasy, amphetamines, cocaine, morphinics).

CONTACTS AND LOCATIONS:
Overall Officials: Aurélie BERGER-VERGIAT, MD, Principal Investigator — Service Addictologie et Psychiatrie des urgences
Locations (1):
- Hôpital Edouard Herriot, Lyon, France